CLINICAL TRIAL: NCT06460519
Title: Prevalence of the Aortic to Radial Pressure Gradient in States of Shock
Brief Title: The Prevalence of the Aortic to Radial Pressure Gradient in States of Shock, Outside the Context of Cardiac Surgery, a Prospective Study
Acronym: PARECHOC
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0264
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-10

CONDITIONS: Shock
Keywords: Radial artery; Femoral artery; Norepinephrine equivalent; Intensive care unit
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intensive care unit patient with shock, who don't be in perioperative of cardiac surgery: Patients of age superior or equal of 18 years, with a vasopressor support superior 0.5 µg/kg/min of equivalent norepinephrine during more than 30 minutes.
  The patients are not in perioperative of cardiac surgery (between the beginning of the intervention and 7 days after).
  The patients have a monitoring of arterial pressure with a radial arterial catheter, and the physician decided to have a monitoring of arterial pressure with a femoral arterial catheter.
  Interventions: Other: Non-invasive blood pressure measurements

INTERVENTIONS:
Other: Non-invasive blood pressure measurements — Non-invasive blood pressure measurements to the tension cuff three times in a row on each side (right arm and left arm)

SUMMARY:
First described in cardiac surgery, the aortic to radial pressure gradient (ATRAP) is the cause of an underestimation of the aortic pressure with a measure assumed with a radial catheter, and he can concert 1 of 3rd patients. The risks factor well known are small height, previous hypertension, long and difficult surgery, radial artery diameter less than 1.8mm.

The ATRAP definition is a pressure difference between radial and femoral (same of the aortic pressure) pressure of 25mmHg on the systolic pressure, or a pressure difference on the mean pressure of 10mmHg, both measures realised by arterial canulation, and with a duration superior than 5 minutes.

If this gradient appears in pathophysiological specifics situations, there is a risk of inappropriate administration of vasopressors, with more hospitalisation days, more side effect of vasopressors like an augmentation of myocardial work.

The ATRAP is documented in septic shock with a prevalence between 21% and 27%. The ATRAP can appear in shocks, moreover with doses of equivalent norepinephrine of 0.5 µg/kg/min who is use for the definition of refractive shock, the difference between the two pressure is higher if the dose of equivalent norepinephrine is higher than 1µg/kg/min. But the prevalence and risks factors are barely unknowns in this situation.

Most of the time, a radial arterial catheter is used for hemodynamic monitoring for his simplicity of utilisation and the lows complications associated. Some medical teams in cardiac surgeries, or in intensive care unit (ICU) for the management of shocks used often radial and femoral arterial catheter. It seems there is no at risk for the utilisation of a radial and femoral arterial canulation.

Out of the situation of cardiac surgery, there is a lack of information of the ATRAP, the objective of the study is to evaluate the prevalence of the ATRAP in shock, out of the situation of cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* age superior or equal 18 years
* Vasopressors support superior or equal 0.5 µg/kg/min of equivalent norepinephrine
* Invasive monitoring of blood pressure with a radial arterial catheter and a femoral arterial catheter decided by de physician
* Beginning of the shock less than 48 hours.
* Consent

Exclusion Criteria:

* perioperative of cardiac surgery (between the beginning of the surgery and 7 days after)
* pregnant woman or breast-feeding
* Major person under protection
* Person with privation of liberty by a justice decision, or an administrative decision

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 180 patients of intensive care unit (ICU), in shock with equal or more than 0.5µg/kg/min of norepinephrine equivalent, who are not in perioperative of cardiac surgery. And who have a monitoring of arterial pressure by a radial catheter, and for who the physician decided to put in place a femoral arterial catheter.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-11-03 (Estimated); Study Completion 2026-11-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence (percentage) of ATRAP is determined by the ratio of patients with ATRAP to total. ATRAP is defined by a 25mmHg systolic or 10mmHg mean pressure difference between radial and femoral arterial pressures during more than 5 minutes. | The primary outcome will be measure at the inclusion of the patient when the femoral arterial catheter will be in place.
  The prevalence of the ATRAP will be show in percentage (%), with his confidence interval at 95%.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Département d'anesthésie Réanimation Hôpital Cardiologique Louis Pradel/Groupement Hospitalier Est, Bron
  - Hopital Edouard heriot/Groupement hospitalier Centre, service de médecine intensive réanimation, Lyon
  - Hôpital Edouard Heriot/ Groupement hospitalier Centre, service d'anesthésie réanimation, Lyon
  - Hôpital de la Croix-Rousse/Groupement hospitalier Nord, service d'anesthésie réanimation, Lyon
  - Centre hospitalier Lyon Sud/Groupement hospitalier Sud, Service d'anesthésie réanimation médecine intensive, Lyon

IPD SHARING:
Plan to Share IPD: No